CLINICAL TRIAL: NCT02838147
Title: Effect of a Continuous Glucose Monitoring on Maternal and Neonatal Outcomes in Gestational Diabetes Mellitus: A Randomized Controlled Trial
Brief Title: Effect of a Continuous Glucose Monitoring on Maternal and Neonatal Outcomes in Gestational Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0213-16- TLV
Record Dates: First submitted 2016-07-17; First posted 2016-07-20 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: GDM

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal OGTT (Oral Glucose Tolerance Test) (Experimental): Patients with normal OGTT (4 normal values) - will be allocated to 2-week period to FreeStyle sensors.
  Interventions: Device: FreeStyle sensors.
- Pathological OGTT - 1 abnormal value (Experimental): Patients will pathological OGTT (either one or more abnormal values) will be randomly allocated to the antenatal care plus FreeStyle group or the SMBG group by a computer generated random number table
  Interventions: Device: FreeStyle sensors.; Device: Glucometer
- Pathological OGTT - 2 abnormal value (Experimental): Patients will pathological OGTT (either one or more abnormal values) will be randomly allocated to the antenatal care plus FreeStyle group or the SMBG group by a computer generated random number table
  Interventions: Device: FreeStyle sensors.; Device: Glucometer

INTERVENTIONS:
Device: FreeStyle sensors. — Patients with normal OGTT (4 normal values) - will be allocated to 2-week period to FreeStyle sensors.
Device: Glucometer — Patients with pathological OGTT - 1 abnormal value Patients with pathological OGTT - 2 abnormal value
  Arms: Pathological OGTT - 1 abnormal value; Pathological OGTT - 2 abnormal value

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as carbohydrate intolerance first diagnosed during pregnancy [1]. It is associated with adverse pregnancy outcome for the mother, and the fetus with consequences regarding future health and development of the neonate. Maternal consequences include increased rate of operative and cesarean delivery, hypertensive disorders during pregnancy and future risk for type 2 diabetes mellitus (T2DM) as well as other aspects of the metabolic syndrome, such as obesity, cardiovascular morbidities and recurrent GDM [2-4]. Also, children born to mothers affected by gestational hypertension have been found to have higher body mass index (BMI), systolic blood pressure, glucose and insulin levels [5]; this risk extends into adulthood, with an 8-fold increased risk of type 2 diabetes among young adults exposed to gestational diabetes during fetal life [6].

Of all types of diabetes, GDM accounts for approximately 90-95% of all cases [4, 7]. It complicates up to 14% of all pregnancies. Its prevalence is increasing and parallels the rising incidence of type 2 diabetes mellitus worldwide [3,4]. Risk factors for developing GDM in pregnancy include obesity, previously GDM, glycosuria, family history, ethnicity and hypertension [5,6].

DETAILED DESCRIPTION:
Introduction

Gestational diabetes mellitus (GDM) is defined as carbohydrate intolerance first diagnosed during pregnancy [1]. It is associated with adverse pregnancy outcome for the mother, and the fetus with consequences regarding future health and development of the neonate. Maternal consequences include increased rate of operative and cesarean delivery, hypertensive disorders during pregnancy and future risk for type 2 diabetes mellitus (T2DM) as well as other aspects of the metabolic syndrome, such as obesity, cardiovascular morbidities and recurrent GDM [2-4]. Also, children born to mothers affected by gestational hypertension have been found to have higher body mass index (BMI), systolic blood pressure, glucose and insulin levels [5]; this risk extends into adulthood, with an 8-fold increased risk of type 2 diabetes among young adults exposed to gestational diabetes during fetal life [6].

Of all types of diabetes, GDM accounts for approximately 90-95% of all cases [4, 7]. It complicates up to 14% of all pregnancies. Its prevalence is increasing and parallels the rising incidence of type 2 diabetes mellitus worldwide [3,4]. Risk factors for developing GDM in pregnancy include obesity, previously GDM, glycosuria, family history, ethnicity and hypertension [5,6].

It has been clearly demonstrated that intensified management and the achievement of established levels of glycemic control using memory-based self-monitoring blood glucose, glyburide treatment or if needed multiple injections of insulin, diet, and an interdisciplinary team effort was associated with enhanced pregnancy outcome [8-10]. The above recommendations support the routine use of self-monitoring blood glucose in the management of the pregnancy compromised by diabetes. The recommendation of the American Colleague of Obstetrics and Gynecology as recently published [11] are four-times daily glucose monitoring preformed as fasting and either 1 or 2 hours after each meal with possible modifications made in diet-controlled GDM patients after reaching well controlled glucose levels.

The role of self-monitoring blood glucose in intensified therapy in non-pregnant and pregnant women has become the standard to achieve targeted levels of glycemic control. Yet, self-monitoring blood glucose may have some disadvantages. It is painful to perform. Another shortcoming in the use of reflectance meters is that each glucose determination represents a sole glucose value during the day, a "snap shot" of glucose value.

Recently, several companies have attempted to develop a new technology that measures continuous glucose. Some of these techniques are non-invasive while others are minimally invasive. Continuous glucose monitoring system (CGMS) employs four different approaches: transdermal, glucose electrode, micro-dialysis or open-flow micro perfusion. Currently, two are commercially available. The transdermal approach (Glucowatch; Cygnus, CA, USA) employs reverse iontophoresis by applying low voltage current to the skin surface causing interstitial fluid (containing glucose) to pass through the skin [12]. Glucose is then measured by an oxidase reaction. This data also contains information about skin temperature and sweat that are all included in the calculation process. The MiniMed CGM System (Sylmar, CA, USA) is composed of a disposable subcutaneous glucose-sensing device and an electrode impregnated with glucose oxidase connected by a cable to a lightweight monitor which is worn over clothing or a belt [13]. The system measures glucose levels every 10 seconds, based on the electrochemical detection of glucose by its reaction with glucose oxidase, and stores an average value every 5 minutes, for a total of 288 measurements per day. The glucose measurement is performed in subcutaneous tissue in which the interstitial glucose levels are in the range of 40-400 mg/dl. The data are stored in the monitor for later downloading and reviewing on a personal computer. The patients are unaware of the results of the sensor measurements during the monitoring period. Glucose values obtained with CGMS have been shown to correlate with laboratory measurements of plasma glucose levels [14] and with home glucose meter values [15].

The CGMS has been studied in non-pregnant patients where it has demonstrated clinical usefulness by enhancing decision-making through detecting previously unrecognized postprandial hyperglycemia and nocturnal hyper-and hypoglycemia [16]. Scientific evidence on a HbA1c-reducing effect of CGMS use is limited [17, 18]. Although some studies do evaluate the effect of CGMS use on biochemical endpoints, such as HbA1c levels, data on clinical endpoints like diabetic complications, are lacking. The usefulness of CGMS use during pregnancy has hardly been evaluated up to now [18].

There are only limited randomized clinical trials assessing the usefulness of CGMS in reducing the rate of diabetes related pregnancy complications with conflicting results [19, 20]. Murphy et al. [19] showed in 71 pregnant women with Type 1 and 2 diabetes mellitus that intermittent (4-6 weeks interval) CGMS resulted in a significant reduction of HbA1C at 32-36 weeks of gestation, lower birth weight, and reduced risk of macrosomia (odds ratio 0.36, 95% confidence interval 0.13 to 0.98, P<0.05) compared to standard antenatal care. However, this study was hampered by small sample size and both study groups differed in composition (e.g. 5 set of twins in the intervention group as opposed to none in the control group). In contrast, a recently published study [20] of 154 pregnant women with preexisting diabetes mellitus randomized to either real time CGM for 6 days at 8,12,21,27 and 33 weeks of gestation or routine care only showed neither an improvement in glycemic control, reflected in similar rates of hypoglycemia events and HbA1C levels, nor a reduction of large for gestational age neonates rate in the CGM group. In a recent study, Wei et al. included a total of 106 women with GDM in gestational weeks 24-28 were randomly allocated to the antenatal care plus CGMS group or the self-monitoring blood glucose group [21]. The authors showed The proportion of GDM women with excessive gestational weight gain was lower in the CGMS group than in the self-monitoring blood glucose (SMBG) group (33.3% vs. 56.4%, P=0.039), and women who initiated CGMS earlier gained less weight (P=0.017). In addition, the investigators showed that the mode of blood glucose monitoring (adjusted OR 2.40; 95% CI 1.030-5.588; P=0.042) was an independent factor for weight gain.

Since obstetric complications in diabetic pregnancies, especially macrosomia and large for gestational age newborn, seem to be related to glycemic control, the investigators hypothesize that the additional use of will reduce adverse pregnancy outcome related to pregnancies complicated with gestational diabetes.

Aims:

This trial evaluates the clinical effectiveness, costs and cost-effectiveness of Continuous glucose monitoring using FreeStyle Freedom Lite CGMS use with the aim to optimize glycemic control and pregnancy outcome of pregnancies diagnosed with GDM relative to standard control methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological glucose tolerance test (GCT) are eligible for the study.
* Women with a singleton pregnancy who were diagnosed with GDM between 24 and 28 weeks' gestation.

Exclusion Criteria:

* Alcohol or substance abuse, pre-gestational diabetes, any hypertensive disorders and chronic diseases requiring medication except for hypothyroidism. Additionally, multiple gestation, known fetal anomaly or chromosomal defects and intrauterine fetal growth restriction (EFW less than the 10th percentile according to local growth charts) will be excluded as well. Written informed consent will be obtained from all study participants.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Neonatal hypoglycemia | 2 weeks.
  Number of Neonatal hypoglycemia(defined as a blood glucose concentration ≤45mg/dL (2.5mmol/L))

SECONDARY OUTCOMES:
Large-for-gestational age (LGA) | 2 weeks
  Number of patients with LGA defined as birth weight above the 90th percentile
Macrosomia | 2 weeks
  Number of patients with Macrosomia defined as birth weight > 4,000g

CONTACTS AND LOCATIONS:
Overall Officials: yariv yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No